CLINICAL TRIAL: NCT07246928
Title: US-guided Intralesional Injection of Cystic Hygroma - A Case Report
Acronym: US: Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Sarah Arafat, Lecturer of Oral and Maxillofacial Surgery, Faculty of Oral and Dental Medicine, Delta University for Science & Technology, Delta University for Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 025091866
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Intralesional Injection of Cystic Hygroma

STUDY DESIGN:
Intervention Model Description: Case Report
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pediatric patient (Experimental)
  Interventions: Procedure: Intralesional Injection of Bleomycin

INTERVENTIONS:
Procedure: Intralesional Injection of Bleomycin — Aspiration of Cystic Hygroma Fluid and Intralesional Injection

SUMMARY:
Ultrasound-guided Intralesional Injection of Cystic Hygroma - A Case Report

DETAILED DESCRIPTION:
Ultrasound-guided Intralesional Injection of Cystic Hygroma [lymphatic malformation]

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients of age up to 12 years having cystic hygromas (macrocystic lymphatic malformations), from the vascular anomalies clinic at the pediatric surgery department in Cairo University Specialized Pediatric Hospital (Abu EL-Reesh hospital). -

Exclusion Criteria:

pediatric patients with lung, liver, or kidney diseases -

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
improvement: reduction in lesion size | one year
  reduction in lesion size
improvement: reduction of lesion size | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gamal El-Tagy, MD, Study Director — pediatric surgery department, Cairo University
Locations (1):
- Specialized Pediatric Hospital (Abu EL-Reesh Japanese hospital), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided